CLINICAL TRIAL: NCT02886832
Title: A Pilot, Open-label Study to Evaluate the Effects of a Prostate Health Formulation on Scores Attained From the International Prostate Symptom Score (I-PSS) Questionnaire Among Overall Healthy Male Participants Who Report Lower Urinary Tract Complaints
Brief Title: A Study to Evaluate the Effects of a Prostate Health Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CL089
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Prostate Health
Keywords: Prostate Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostate Health formulation (Experimental): Prostate Health formulation
  Interventions: Dietary Supplement: Prostate Health formulation

INTERVENTIONS:
Dietary Supplement: Prostate Health formulation

SUMMARY:
The purpose of this study is to assess the efficacy of a Prostate Health formulation on scores attained from the I-PSS questionnaire. Safety and tolerability of the formulation will also be assessed.

DETAILED DESCRIPTION:
This study is a pilot, open-label study to evaluate the efficacy, safety and tolerability of a Prostate Health formulation. Each subject will receive a specific dose of the formulation once daily.

Participants will undergo assessments of blood tests, vital signs, body weight, BMI with completion of questionnaires.

The primary objective of the study is to assess effectiveness of the Prostate Health formulation on the I-PSS score.

Secondary objectives:

1. To assess the I-PSS "Quality of Life" question score
2. To assess the PSA level
3. To assess the IIEF-5 questionnaire score
4. To assess body weight
5. To assess BMI
6. To assess the score on a questionnaire for health-related quality of life

ELIGIBILITY:
Primary Inclusion Criteria:

1. Ambulatory, male, 45-75 years of age
2. Having a BMI of 20-35
3. Having an I-PSS score of 1-7
4. Overall healthy and having no difficulty with digestion or absorption of food

Primary Exclusion Criteria:

1. Unable to maintain stable exercise and dietary habits throughout the study
2. History of any of the following medical condition(s): diabetes, prostate and/or bladder cancer, arrhythmia, hypotension, hypertension (unless on a stable dose of anti-hypertensive medication for 3 months prior to Baseline/screening and not likely to change medication or dose during the study period), chronic inflammatory or autoimmune disease, gastrointestinal disease (including gastroesophageal reflux and peptic ulcer), biliary obstruction (past or present), cardiovascular disease, hyper- or hypothyroidism (unless on a stable dose of medication for 3 months prior to Baseline/screening and not likely to change medication or dose during the study period), liver or kidney disease, edema with or without congestive heart failure, stroke, bleeding disorders, sleep apnea, insomnia, migraine headaches (within 3 months prior to Baseline/screening), psychiatric disorders, anxiety disorder, known or suspected estrogen-dependent neoplasia, history of thrombosis or embolism, any neurological disorder that could yield cognitive deterioration including Parkinson's disease, stroke, intracranial hemorrhage, head injury, brain tumor(s), normal pressure hydrocephalus or evidence of delirium, confusion, dementia or Alzheimer's disease, or other condition(s) that would preclude participation in the study in the judgment of the PI/Sub-Investigator (Sub-I)
3. Having taken a 5-alpha-reductase inhibitor, alpha- or beta-blocker medication, diuretics, calcium channel blockers, tricyclic antidepressants, or anticholinergic agents 90 days prior to Baseline/screening
4. Having taken testosterone replacement therapy for less than 3 months or unlikely to maintain the same therapeutic regimen (including dose) throughout the study period
5. Having taken pygeum extract, beta-sitosterol, melatonin, lycopene, or boron and unwilling to discontinue use 30 days prior to enrollment (unless permitted to enroll in the judgment of the PI/Sub-I)
6. Having taken saw palmetto, grass pollen extract, flower pollen extract, stinging and dwarf nettle extract, pumpkin seed oil extract, lignan extract, or boswellia serrata extract less than 6 months prior to screening and unwilling to discontinue use 30 days prior to enrollment (unless permitted to enroll in the judgment of the PI/Sub-I)
7. Currently consuming a product containing olestra and unwilling to discontinue use 30 days prior to enrollment
8. Having taken anxiolytics and sedative hypnotics, anticonvulsants, antineoplastics, anti-migraine medication(s), opioid analgesics, monoamine oxidase inhibitors (MAOIs), phosphodiesterase inhibitors, adenosine reuptake inhibitors, dopamine agonists, dopamine antagonists, or immunosuppressants within 30 days prior to Baseline/screening
9. Having taken an anti-inflammatory medication, antihistamine or decongestant within 14 days prior to Baseline/screening
10. Having had a surgical procedure, including prostate or bladder surgery, which would preclude study participation in the judgment of the PI/Sub-I
11. Having any blood coagulation disorder, anemia, vitamin K deficiency, or taking anticoagulant and antiplatelet medication(s)
12. Having abnormal screening laboratory test values: bilirubin > 2.5 x ULN, AST/SGOT and ALT/SGPT > 2.5 x ULN, serum creatinine > 1.5 mg/dL, PSA > 4 ng/mL, abnormal urinalysis (positive proteins, leukocyte, occult blood and nitrites) or any other lab test result(s) that would preclude study participation in the judgment of the PI/Sub-I
13. Currently consumes more than 6 standard alcoholic drinks per week (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
14. Unable or unwilling to abstain from consuming any alcoholic drink within two hours of taking the study product
15. History of known alcohol or substance abuse (eg, opiates, benzodiazepines, or amphetamines)
16. Having smoked any cigarette, electronic cigarette, cigar, pipe, or recreational drug in the past 30 days
17. History of allergy or sensitivity to any component of the study product (as well as pine)
18. Participation in another study within 30 days prior to Baseline/screening
19. Unable or unwilling to avoid consuming grapefruit
20. Having a pacemaker or any internal medical device

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09-21 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Mean change on I-PSS score | 60 days

SECONDARY OUTCOMES:
Mean change on the I-PSS Quality of Life question score | 60 days
Mean change in the PSA level | 60 days
Mean change on the IIEF-5 questionnaire score | 60 days
Mean change in body weight | 60 days
Mean change in BMI | 60 days
Mean change in the score on a questionnaire for health-related quality of life | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joyal, M.D., Principal Investigator — Life Extension
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adjakly M, Ngollo M, Dagdemir A, Judes G, Pajon A, Karsli-Ceppioglu S, Penault-Llorca F, Boiteux JP, Bignon YJ, Guy L, Bernard-Gallon D. Prostate cancer: The main risk and protective factors-Epigenetic modifications. Ann Endocrinol (Paris). 2015 Feb;76(1):25-41. doi: 10.1016/j.ando.2014.09.001. Epub 2015 Jan 13. PMID 25592466
- [Background] Aguilar F, Autrup H, Barlow S et al. Scientific Opinion of the Panel onf Food Additives, Flavourings, Processing Adids and Materials in Contact with Food on a request from the Commission on the safety in use of lycopene as a food colour. The EFSA Journal. 2008;675:1-66.
- [Background] Andersen LP, Gogenur I, Rosenberg J, Reiter RJ. The Safety of Melatonin in Humans. Clin Drug Investig. 2016 Mar;36(3):169-75. doi: 10.1007/s40261-015-0368-5. PMID 26692007
- [Background] Andro M, Riffaud J. Pygeum Africanum extract for the treatment of patients with benign prostatic hyperplasia: A review of 25 years of published experience. Current Therapeutic Research. 1995;56(8):796-817.
- [Background] Ansari MS, Gupta NP. Lycopene: a novel drug therapy in hormone refractory metastatic prostate cancer. Urol Oncol. 2004 Sep-Oct;22(5):415-20. doi: 10.1016/j.urolonc.2004.05.009. PMID 15464923
- [Background] Assar EA, Vidalle MC, Chopra M, Hafizi S. Lycopene acts through inhibition of IkappaB kinase to suppress NF-kappaB signaling in human prostate and breast cancer cells. Tumour Biol. 2016 Jul;37(7):9375-85. doi: 10.1007/s13277-016-4798-3. Epub 2016 Jan 16. PMID 26779636
- [Background] Awad AB, Chen YC, Fink CS, Hennessey T. beta-Sitosterol inhibits HT-29 human colon cancer cell growth and alters membrane lipids. Anticancer Res. 1996 Sep-Oct;16(5A):2797-804. PMID 8917388
- [Background] Awad AB, Chinnam M, Fink CS, Bradford PG. beta-Sitosterol activates Fas signaling in human breast cancer cells. Phytomedicine. 2007 Nov;14(11):747-54. doi: 10.1016/j.phymed.2007.01.003. Epub 2007 Mar 12. PMID 17350814
- [Background] Awad AB, Gan Y, Fink CS. Effect of beta-sitosterol, a plant sterol, on growth, protein phosphatase 2A, and phospholipase D in LNCaP cells. Nutr Cancer. 2000;36(1):74-8. doi: 10.1207/S15327914NC3601_11. PMID 10798219
- [Background] Awad AB, Roy R, Fink CS. Beta-sitosterol, a plant sterol, induces apoptosis and activates key caspases in MDA-MB-231 human breast cancer cells. Oncol Rep. 2003 Mar-Apr;10(2):497-500. PMID 12579296
- [Background] Azimi H, Khakshur AA, Aghdasi I, Fallah-Tafti M, Abdollahi M. A review of animal and human studies for management of benign prostatic hyperplasia with natural products: perspective of new pharmacological agents. Inflamm Allergy Drug Targets. 2012 Jun;11(3):207-21. doi: 10.2174/187152812800392715. PMID 22512478
- [Background] Barlet A, Albrecht J, Aubert A, Fischer M, Grof F, Grothuesmann HG, Masson JC, Mazeman E, Mermon R, Reichelt H, et al. [Efficacy of Pygeum africanum extract in the medical therapy of urination disorders due to benign prostatic hyperplasia: evaluation of objective and subjective parameters. A placebo-controlled double-blind multicenter study]. Wien Klin Wochenschr. 1990 Nov 23;102(22):667-73. German. PMID 1702916
- [Background] Barranco WT, Eckhert CD. Boric acid inhibits human prostate cancer cell proliferation. Cancer Lett. 2004 Dec 8;216(1):21-9. doi: 10.1016/j.canlet.2004.06.001. PMID 15500945
- [Background] Barranco WT, Eckhert CD. Cellular changes in boric acid-treated DU-145 prostate cancer cells. Br J Cancer. 2006 Mar 27;94(6):884-90. doi: 10.1038/sj.bjc.6603009. PMID 16495920
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Berges RR, Windeler J, Trampisch HJ, Senge T. Randomised, placebo-controlled, double-blind clinical trial of beta-sitosterol in patients with benign prostatic hyperplasia. Beta-sitosterol Study Group. Lancet. 1995 Jun 17;345(8964):1529-32. doi: 10.1016/s0140-6736(95)91085-9. PMID 7540705
- [Background] Bolt HM, Basaran N, Duydu Y. Human environmental and occupational exposures to boric acid: reconciliation with experimental reproductive toxicity data. J Toxicol Environ Health A. 2012;75(8-10):508-14. doi: 10.1080/15287394.2012.675301. PMID 22686310
- [Background] Breza J, Dzurny O, Borowka A, Hanus T, Petrik R, Blane G, Chadha-Boreham H. Efficacy and acceptability of tadenan (Pygeum africanum extract) in the treatment of benign prostatic hyperplasia (BPH): a multicentre trial in central Europe. Curr Med Res Opin. 1998;14(3):127-39. doi: 10.1185/03007999809113352. PMID 9787978
- [Background] Buscemi N, Vandermeer B, Hooton N, Pandya R, Tjosvold L, Hartling L, Vohra S, Klassen TP, Baker G. Efficacy and safety of exogenous melatonin for secondary sleep disorders and sleep disorders accompanying sleep restriction: meta-analysis. BMJ. 2006 Feb 18;332(7538):385-93. doi: 10.1136/bmj.38731.532766.F6. Epub 2006 Feb 10. PMID 16473858
- [Background] Chatelain C, Autet W, Brackman F. Comparison of once and twice daily dosage forms of Pygeum africanum extract in patients with benign prostatic hyperplasia: a randomized, double-blind study, with long-term open label extension. Urology. 1999 Sep;54(3):473-8. doi: 10.1016/s0090-4295(99)00147-8. PMID 10475357
- [Background] Chen P, Zhang W, Wang X, Zhao K, Negi DS, Zhuo L, Qi M, Wang X, Zhang X. Lycopene and Risk of Prostate Cancer: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2015 Aug;94(33):e1260. doi: 10.1097/MD.0000000000001260. PMID 26287411
- [Background] Cui Y, Winton MI, Zhang ZF, Rainey C, Marshall J, De Kernion JB, Eckhert CD. Dietary boron intake and prostate cancer risk. Oncol Rep. 2004 Apr;11(4):887-92. PMID 15010890
- [Background] Culver B, Hubbard S. 1996. Inorganic boron health effects in humans: An aid to risk assessment and clinical judgment. J Trace Elem Exp Med 9:175-184.
- [Background] Devaraj S, Mathur S, Basu A, Aung HH, Vasu VT, Meyers S, Jialal I. A dose-response study on the effects of purified lycopene supplementation on biomarkers of oxidative stress. J Am Coll Nutr. 2008 Apr;27(2):267-73. doi: 10.1080/07315724.2008.10719699. PMID 18689558
- [Background] DHHS. U. S. Department of Health and Human Services. Center for Drug Evaluation and Research. Guidance for Industry. Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapetuics in Adult Heathy Volunteers. 7/2005. http://www.fda.gov/downloads/Drugs/Guidances/UCM078932.pdf. Accessed 6/21/2016.
- [Background] Drake MJ, Mills IW, Noble JG. Melatonin pharmacotherapy for nocturia in men with benign prostatic enlargement. J Urol. 2004 Mar;171(3):1199-202. doi: 10.1097/01.ju.0000110442.47593.ea. PMID 14767300
- [Background] Gallardo-Williams MT, Chapin RE, King PE, Moser GJ, Goldsworthy TL, Morrison JP, Maronpot RR. Boron supplementation inhibits the growth and local expression of IGF-1 in human prostate adenocarcinoma (LNCaP) tumors in nude mice. Toxicol Pathol. 2004 Jan-Feb;32(1):73-8. doi: 10.1080/01926230490260899. PMID 14713551
- [Background] Gooneratne NS, Edwards AY, Zhou C, Cuellar N, Grandner MA, Barrett JS. Melatonin pharmacokinetics following two different oral surge-sustained release doses in older adults. J Pineal Res. 2012 May;52(4):437-45. doi: 10.1111/j.1600-079X.2011.00958.x. Epub 2012 Feb 21. PMID 22348451
- [Background] Grattan BJ Jr. Plant sterols as anticancer nutrients: evidence for their role in breast cancer. Nutrients. 2013 Jan 31;5(2):359-87. doi: 10.3390/nu5020359. PMID 23434903
- [Background] Gupta R, Sharma AK, Dobhal MP, Sharma MC, Gupta RS. Antidiabetic and antioxidant potential of beta-sitosterol in streptozotocin-induced experimental hyperglycemia. J Diabetes. 2011 Mar;3(1):29-37. doi: 10.1111/j.1753-0407.2010.00107.x. PMID 21143769
- [Background] Hansen MV, Andersen LT, Madsen MT, Hageman I, Rasmussen LS, Bokmand S, Rosenberg J, Gogenur I. Effect of melatonin on depressive symptoms and anxiety in patients undergoing breast cancer surgery: a randomized, double-blind, placebo-controlled trial. Breast Cancer Res Treat. 2014 Jun;145(3):683-95. doi: 10.1007/s10549-014-2962-2. Epub 2014 Apr 23. PMID 24756186
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Heber D, Lu QY. Overview of mechanisms of action of lycopene. Exp Biol Med (Maywood). 2002 Nov;227(10):920-3. doi: 10.1177/153537020222701013. PMID 12424335
- [Background] Heindel JJ, Price CJ, Field EA, Marr MC, Myers CB, Morrissey RE, Schwetz BA. Developmental toxicity of boric acid in mice and rats. Fundam Appl Toxicol. 1992 Feb;18(2):266-77. doi: 10.1016/0272-0590(92)90055-m. PMID 1601227
- [Background] Henderson K, Stella SL, Kobylewski S, Eckhert CD. Receptor activated Ca(2+) release is inhibited by boric acid in prostate cancer cells. PLoS One. 2009 Jun 23;4(6):e6009. doi: 10.1371/journal.pone.0006009. PMID 19554099
- [Background] Hendriks HF, Brink EJ, Meijer GW, Princen HM, Ntanios FY. Safety of long-term consumption of plant sterol esters-enriched spread. Eur J Clin Nutr. 2003 May;57(5):681-92. doi: 10.1038/sj.ejcn.1601598. PMID 12771969
- [Background] Hevia D, Gonzalez-Menendez P, Quiros-Gonzalez I, Miar A, Rodriguez-Garcia A, Tan DX, Reiter RJ, Mayo JC, Sainz RM. Melatonin uptake through glucose transporters: a new target for melatonin inhibition of cancer. J Pineal Res. 2015 Mar;58(2):234-50. doi: 10.1111/jpi.12210. Epub 2015 Feb 7. PMID 25612238
- [Background] Ilic D. Lycopene for the prevention and treatment of prostate disease. Recent Results Cancer Res. 2014;202:109-14. doi: 10.1007/978-3-642-45195-9_13. PMID 24531784
- [Background] Jahnke G, Marr M, Myers C, Wilson R, Travlos G, Price C. Maternal and developmental toxicity evaluation of melatonin administered orally to pregnant Sprague-Dawley rats. Toxicol Sci. 1999 Aug;50(2):271-9. doi: 10.1093/toxsci/50.2.271. PMID 10478864
- [Background] Jian L, Du CJ, Lee AH, Binns CW. Do dietary lycopene and other carotenoids protect against prostate cancer? Int J Cancer. 2005 Mar 1;113(6):1010-4. doi: 10.1002/ijc.20667. PMID 15514967
- [Background] Jung-Hynes B, Huang W, Reiter RJ, Ahmad N. Melatonin resynchronizes dysregulated circadian rhythm circuitry in human prostate cancer cells. J Pineal Res. 2010 Aug;49(1):60-8. doi: 10.1111/j.1600-079X.2010.00767.x. Epub 2010 May 27. PMID 20524973
- [Background] Jung-Hynes B, Schmit TL, Reagan-Shaw SR, Siddiqui IA, Mukhtar H, Ahmad N. Melatonin, a novel Sirt1 inhibitor, imparts antiproliferative effects against prostate cancer in vitro in culture and in vivo in TRAMP model. J Pineal Res. 2011 Mar;50(2):140-9. doi: 10.1111/j.1600-079X.2010.00823.x. Epub 2010 Nov 9. PMID 21062352
- [Background] Kava. In: Natural Medicines Comprehensive Database. Stockton, CA: Therapeutic Research Faculty. [Updated January 6, 2016; Accessed May 24, 2016]. http://naturaldatabase.therapeuticresearch.com/nd/Search.aspx?cs=OSU&s=ND&pt=100&id=872&ds =&name=KAVA&searchid=37784702
- [Background] Kim CH, Yoo YM. Melatonin Induces Apoptotic Cell Death via p53 in LNCaP Cells. Korean J Physiol Pharmacol. 2010 Dec;14(6):365-9. doi: 10.4196/kjpp.2010.14.6.365. Epub 2010 Dec 31. PMID 21311676
- [Background] Klippel KF, Hiltl DM, Schipp B. A multicentric, placebo-controlled, double-blind clinical trial of beta-sitosterol (phytosterol) for the treatment of benign prostatic hyperplasia. German BPH-Phyto Study group. Br J Urol. 1997 Sep;80(3):427-32. PMID 9313662
- [Background] Kucuk O, Sarkar FH, Djuric Z, Sakr W, Pollak MN, Khachik F, Banerjee M, Bertram JS, Wood DP Jr. Effects of lycopene supplementation in patients with localized prostate cancer. Exp Biol Med (Maywood). 2002 Nov;227(10):881-5. doi: 10.1177/153537020222701007. PMID 12424329
- [Background] Larre S, Camparo P, Comperat E, Boulbes D, Haddoum M, Baulande S, Soularue P, Costa P, Cussenot O. Biological effect of human serum collected before and after oral intake of Pygeum africanum on various benign prostate cell cultures. Asian J Androl. 2012 May;14(3):499-504. doi: 10.1038/aja.2011.132. Epub 2011 Dec 26. PMID 22198631
- [Background] Lee WH, Isaacs WB, Bova GS, Nelson WG. CG island methylation changes near the GSTP1 gene in prostatic carcinoma cells detected using the polymerase chain reaction: a new prostate cancer biomarker. Cancer Epidemiol Biomarkers Prev. 1997 Jun;6(6):443-50. PMID 9184779
- [Background] Levin RM, Das AK. A scientific basis for the therapeutic effects of Pygeum africanum and Serenoa repens. Urol Res. 2000 Jun;28(3):201-9. doi: 10.1007/s002409900098. PMID 10929430
- [Background] Li D, Chen L, Zhao W, Hao J, An R. MicroRNA-let-7f-1 is induced by lycopene and inhibits cell proliferation and triggers apoptosis in prostate cancer. Mol Med Rep. 2016 Mar;13(3):2708-14. doi: 10.3892/mmr.2016.4841. Epub 2016 Feb 2. PMID 26847233
- [Background] Litovitz TL, Klein-Schwartz W, Oderda GM, Schmitz BF. Clinical manifestations of toxicity in a series of 784 boric acid ingestions. Am J Emerg Med. 1988 May;6(3):209-13. doi: 10.1016/0735-6757(88)90001-0. PMID 3370093
- [Background] Lomenick B, Shi H, Huang J, Chen C. Identification and characterization of beta-sitosterol target proteins. Bioorg Med Chem Lett. 2015 Nov 1;25(21):4976-4979. doi: 10.1016/j.bmcl.2015.03.007. Epub 2015 Mar 11. PMID 25804720
- [Background] Mace, A.E. (1964), Sample Size Determination, New York: Reinhold Publishing Corporation
- [Background] Murray FJ. A comparative review of the pharmacokinetics of boric acid in rodents and humans. Biol Trace Elem Res. 1998 Winter;66(1-3):331-41. doi: 10.1007/BF02783146. PMID 10050928
- [Background] Murray FJ. A human health risk assessment of boron (boric acid and borax) in drinking water. Regul Toxicol Pharmacol. 1995 Dec;22(3):221-30. doi: 10.1006/rtph.1995.0004. PMID 8837846
- [Background] Paroni R, Terraneo L, Bonomini F, Finati E, Virgili E, Bianciardi P, Favero G, Fraschini F, Reiter RJ, Rezzani R, Samaja M. Antitumour activity of melatonin in a mouse model of human prostate cancer: relationship with hypoxia signalling. J Pineal Res. 2014 Aug;57(1):43-52. doi: 10.1111/jpi.12142. Epub 2014 May 20. PMID 24786921
- [Background] Pizzorno L. Nothing Boring About Boron. Integr Med (Encinitas). 2015 Aug;14(4):35-48. PMID 26770156
- [Background] Quiles MT, Arbos MA, Fraga A, de Torres IM, Reventos J, Morote J. Antiproliferative and apoptotic effects of the herbal agent Pygeum africanum on cultured prostate stromal cells from patients with benign prostatic hyperplasia (BPH). Prostate. 2010 Jul 1;70(10):1044-53. doi: 10.1002/pros.21138. PMID 20503393
- [Background] Reagan-Shaw S, Nihal M, Ahmad N. Dose translation from animal to human studies revisited. FASEB J. 2008 Mar;22(3):659-61. doi: 10.1096/fj.07-9574LSF. Epub 2007 Oct 17. PMID 17942826
- [Background] Risk Profile. Beta-sitosterol. CAS No. 83-46-5. http://www.mattilsynet.no/kosmetikk/stoffer_i_kosmetikk/risk_profile_betasitosterol.11370/binary/Risk%20Profile%20Beta-Sitosterol. 8/27/2012. Accessed 6/20/2016.
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462
- [Background] Sainz RM, Mayo JC, Tan DX, Leon J, Manchester L, Reiter RJ. Melatonin reduces prostate cancer cell growth leading to neuroendocrine differentiation via a receptor and PKA independent mechanism. Prostate. 2005 Apr 1;63(1):29-43. doi: 10.1002/pros.20155. PMID 15378522
- [Background] Schwarz S, Obermuller-Jevic UC, Hellmis E, Koch W, Jacobi G, Biesalski HK. Lycopene inhibits disease progression in patients with benign prostate hyperplasia. J Nutr. 2008 Jan;138(1):49-53. doi: 10.1093/jn/138.1.49. PMID 18156403
- [Background] Shao A, Hathcock JN. Risk assessment for the carotenoids lutein and lycopene. Regul Toxicol Pharmacol. 2006 Aug;45(3):289-98. doi: 10.1016/j.yrtph.2006.05.007. Epub 2006 Jun 30. PMID 16814439
- [Background] Shenouda NS, Sakla MS, Newton LG, Besch-Williford C, Greenberg NM, MacDonald RS, Lubahn DB. Phytosterol Pygeum africanum regulates prostate cancer in vitro and in vivo. Endocrine. 2007 Feb;31(1):72-81. doi: 10.1007/s12020-007-0014-y. PMID 17709901
- [Background] Sohn EJ, Won G, Lee J, Lee S, Kim SH. Upregulation of miRNA3195 and miRNA374b Mediates the Anti-Angiogenic Properties of Melatonin in Hypoxic PC-3 Prostate Cancer Cells. J Cancer. 2015 Jan 1;6(1):19-28. doi: 10.7150/jca.9591. eCollection 2015. PMID 25553085
- [Background] Srinivasan V, Pandi-Perumal SR, Brzezinski A, Bhatnagar KP, Cardinali DP. Melatonin, immune function and cancer. Recent Pat Endocr Metab Immune Drug Discov. 2011 May;5(2):109-23. doi: 10.2174/187221411799015408. PMID 22074586
- [Background] Stokinger HE. 1981. The halogens and nonmetals boron and silicon. In: Clayton GD, Clayton FE, eds. Patty's Industrial Hygiene and Toxicology, Vol. 2B. New York: John Wiley and Sons. Pp. 2978- 3005.
- [Background] Sugaya K, Nishijima S, Miyazato M, Kadekawa K, Ogawa Y. Effects of melatonin and rilmazafone on nocturia in the elderly. J Int Med Res. 2007 Sep-Oct;35(5):685-91. doi: 10.1177/147323000703500513. PMID 17900408
- [Background] Ulbricht CE. An Evidence-Based Systematic Review of Beta-Sitosterol, Sitosterol (22,23- dihydrostigmasterol, 24-ethylcholesterol) by the Natural Standard Research Collaboration. J Diet Suppl. 2016;13(1):35-92. Epub 2015 Aug 13. PMID 26268617
- [Background] von Holtz RL, Fink CS, Awad AB. beta-Sitosterol activates the sphingomyelin cycle and induces apoptosis in LNCaP human prostate cancer cells. Nutr Cancer. 1998;32(1):8-12. doi: 10.1080/01635589809514709. PMID 9824850
- [Background] Wade AG, Farmer M, Harari G, Fund N, Laudon M, Nir T, Frydman-Marom A, Zisapel N. Add-on prolonged-release melatonin for cognitive function and sleep in mild to moderate Alzheimer's disease: a 6-month, randomized, placebo-controlled, multicenter trial. Clin Interv Aging. 2014 Jun 18;9:947-61. doi: 10.2147/CIA.S65625. eCollection 2014. PMID 24971004
- [Background] Wang Y, Jacobs EJ, Newton CC, McCullough ML. Lycopene, tomato products and prostate cancer-specific mortality among men diagnosed with nonmetastatic prostate cancer in the Cancer Prevention Study II Nutrition Cohort. Int J Cancer. 2016 Jun 15;138(12):2846-55. doi: 10.1002/ijc.30027. Epub 2016 Feb 23. PMID 26830232
- [Background] Wertz K. Lycopene effects contributing to prostate health. Nutr Cancer. 2009;61(6):775-83. doi: 10.1080/01635580903285023. PMID 20155615
- [Background] Wertz K, Siler U, Goralczyk R. Lycopene: modes of action to promote prostate health. Arch Biochem Biophys. 2004 Oct 1;430(1):127-34. doi: 10.1016/j.abb.2004.04.023. PMID 15325920
- [Background] Wilt T, Ishani A, Mac Donald R, Rutks I, Stark G. Pygeum africanum for benign prostatic hyperplasia. Cochrane Database Syst Rev. 2002;1998(1):CD001044. doi: 10.1002/14651858.CD001044. PMID 11869585
- [Background] Wilt TJ, MacDonald R, Ishani A. beta-sitosterol for the treatment of benign prostatic hyperplasia: a systematic review. BJU Int. 1999 Jun;83(9):976-83. doi: 10.1046/j.1464-410x.1999.00026.x. PMID 10368239
- [Background] Wu K, Erdman JW Jr, Schwartz SJ, Platz EA, Leitzmann M, Clinton SK, DeGroff V, Willett WC, Giovannucci E. Plasma and dietary carotenoids, and the risk of prostate cancer: a nested case-control study. Cancer Epidemiol Biomarkers Prev. 2004 Feb;13(2):260-9. doi: 10.1158/1055-9965.epi-03-0012. PMID 14973107
- [Background] Zhao Y, Chang SK, Qu G, Li T, Cui H. Beta-sitosterol inhibits cell growth and induces apoptosis in SGC-7901 human stomach cancer cells. J Agric Food Chem. 2009 Jun 24;57(12):5211-8. doi: 10.1021/jf803878n. PMID 19456133
- [Derived] Hirsh SP, Pons M, Joyal SV, Swick AG. Self-Assessed Benefits of a Prostate Health Formulation on Nocturia in Healthy Males With Mild Lower Urinary Tract Symptoms: An Open Label Study. Glob Adv Health Med. 2020 Nov 27;9:2164956120973639. doi: 10.1177/2164956120973639. eCollection 2020. PMID 33294303